CLINICAL TRIAL: NCT02469168
Title: Epidermal Coverage of Traumatic Wound Injuries Via Use of Autologous Skin Cell Harvesting Device in Combination With Widened Meshed Autograft Applied Over Bilayered Wound Matrix
Brief Title: Epidermal Coverage of Traumatic Wound Injuries Via Use of Autologous Spray Skin Applied Over Bilayered Wound Matrix
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Rubin, J. Peter, MD (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Leon Nesti, Associate Professor, Walter Reed National Military Medical Center
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WRNNMC 391911-5
Record Dates: First submitted 2015-06-03; First posted 2015-06-11 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Wounds and Injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ReCell (Experimental): Allocation of treatments (Recell vs Control) to the INTEGRA™ Meshed Bilayer Wound Matrix (MBWM). Each patient serves as their own control. Their study treatment area will be divided into Area A and Area B. Investigational treatment will be randomly allocated to either Area A or Area B
  Interventions: Device: Recell
- Control (Active Comparator): Allocation of treatments (Recell vs Control) to the INTEGRA™ Meshed Bilayer Wound Matrix (MBWM). Each patient serves as their own control. Their study treatment area will be divided into Area A and Area B. Investigational treatment will be randomly allocated to either Area A or Area B
  Interventions: Procedure: Control

INTERVENTIONS:
Device: Recell — ReCell Treatment over wound pretreated with INTEGRA™ MBWM Wound Matrix
  Arms: ReCell
Procedure: Control — Standard meshed split thickness skin graft over wound pretreated with INTEGRA™ MBWM Wound Matrix
  Arms: Control

SUMMARY:
The purpose of this investigation is to evaluate the safety, tolerability, preliminary and long-term effectiveness of utilizing the ReCell Autologous Cell Harvesting Device (ReCell) combined with widened split-thickness skin graft (STSG) mesh onto the dermal regenerate INTEGRA™ Meshed Bilayer Wound Matrix (MBWM) for healing of full-thickness wounds.

DETAILED DESCRIPTION:
The goal of the study described herein is to determine the safety, tolerability, preliminary and long-term effectiveness of the use of the Recell device over a widened STSG mesh. It is hypothesized the ReCell cell suspension, in combination with INTEGRA™ MBWM, will improve upon the current standard of care. The potential for ReCell's promotion of healing in the interstices of the STSG mesh may close gaps that are potential points of failure during subsequent rehabilitation and return to physical activity. Within the current study, each participant will serve as his/her own control, allowing for comparison of ReCell treated (experimental) and non-ReCell treated (control) regions of the grafted wound. In the proposed study, each patient will serve as his/her own control. Due to the nature of the study, only patients whose wounds have been previously successfully treated with INTEGRA™ MBWM as part of their standard of care will qualify for participation.

Therefore, as part of enrollment eligibility criteria for this study, the identified study wound will first be treated with INTEGRA™ MBWM. The wound will then be allowed to heal for approximately two to four weeks, at which time a viable granulation layer will have developed thus allowing for next stage STSG grafting. The timing of the STSG application will be determined by clinician judgment based on the state of the granulation process, which varies between patients, but typically takes 2 to 4 weeks.

Approximately two to four weeks after INTEGRA™ MBWM treatment, the studied wound will be divided into a ReCell-treated area (over 1:5 meshed STSG) and a control area treated with 1:1.5 meshed STSG (no ReCell). In all cases, the ReCell region may be up to 320cm2 in size; the upper limit of application area for one ReCell kit, with a similarly sized control region. If the wound is larger than the combined ReCell and control regions (over 640cm2), the areas outside the study regions will be designated as non-study areas and treated according to standard of care. The same primary and secondary dressings will be used on ReCell-treated areas, control areas and donor sites. Once the study and control wounds are determined to have healed, standard local clinical practice will be followed.

Within-subject comparisons of the ReCell region and control region, in order to evaluate improvements associated with use of ReCell, a battery of measurements and evaluations will be made. These measurements are divided into three categories: safety and tolerability, preliminary effectiveness (acute healing process) and long-term effectiveness.

The safety of research participants is foremost. Therefore, efforts will be made to control risks to participants throughout the duration of their study participation. Wound healing time, donor site morbidity and histology will be assessed during an acute 6 week phase, with follow-up visits at Weeks 1, 2, 3, 4 and 6 post-treatment.

Subjects will continue in the study for long-term follow-up with clinic visits at Week 12 and 24 post-treatment. Healing of treated wound sites (A region and B region) and donor sites (STSG 1:5, STSG 1:1.5 and ReCell) will be assessed at each visit. Treated wounds will be considered healed when 95% or greater of the study area has re-epithelialized by Week 6 post-treatment. Donor sites will be considered healed when ≥95% of the donor site has re-epithelialized by Week 4 post-treatment. Aesthetic and functional outcomes of the treated areas will be assessed and documented. Subject satisfaction will also be assessed and documented at these two time points.

ELIGIBILITY:
Inclusion Criteria:

* • The subject is a male or female military healthcare beneficiary of any race or ethnicity, aged 18 years or older, who is being treated for a traumatic wound at WRNMMC

  * The subject has soft tissue loss resulting from a traumatic mechanism such as an explosive blast (i.e. motar, rocket, IED), high-velocity shells (i.e. missile), an avulsion injury, gunshot wound motor vehicle accident and/or burn secondary to blast
  * The subject's full-thickness or deep partial-thickness traumatic wound injury has been treated with INTEGRA™ MBWM as part of their standard of care
  * The wound area is at least 200 cm2
  * All areas of the study wound area are covered with INTEGRA™ MBWM and has fully engrafted - engrafting defined as the presence of a contiguous vascularized granulation layer indicated by the formation of a viable granulation layer (Note: there may be some areas of incomplete granulation at the INTEGRA™ MBWM application site, these areas will be excluded from the study wound area).
  * The subject will comply with protocol requirements
  * The subject will provide voluntary written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization

Exclusion Criteria:

* Subjects will not be eligible for study participation if they meet any of the following criteria:

  * The subject is pregnant and/or lactating (self-reported)
  * The subject has evidence of the following lab value results:

    1. Hematocrit ≤ 20%
    2. INR > 1.8 second
    3. Creatinine (serum) > 2.0 mg/dL
    4. Bilirubin Total (serum) within upper limit of normal (normal range 0.3-1.9 md/dL
    5. Liver function test (AST/ALT) greater than 2 times upper limit of normal as defined by the clinical laboratory defined normal ranges
    6. Albumin (serum) < 2.0 g/dL
    7. Platelets < 70 K/µL
  * The subject's targeted traumatic wound injury is a craniofacial wound
  * The subject's targeted traumatic wound injury is on a weight-bearing surface
  * The subject's targeted traumatic wound is a full-thickness burn injury with visible eschar present (Note: Subjects with a traumatic wound of a burn nature secondary to an explosive blast injury resulting in significant soft tissue loss will NOT be excluded)
  * The subject has active infection processes, that in the opinion of the investigator may compromise safety or study objectives
  * The subject is known to have a pre-existing condition that may interfere with wound healing, e.g. malignancy, diabetes or autoimmune disease, immunocompromised blood borne diseases, has AIDS, is HIV or Hepatitis-A positive, or currently has a severe dermatological disorder (e.g. severe psoriasis, epidermolysis bullosa, pyoderma gangrenosum)
  * The subject has other concurrent conditions that in the opinion of the investigator may compromise safety or study objectives
  * The subject has a known hypersensitivity to Trypsin and/or Compound Sodium Lactate for Irrigation (Hartmann's) solution
  * The subject cannot be compliant with study procedures and that, in the investigator's opinion, would interfere with the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon J Nesti, PhD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Moiemen NS, Vlachou E, Staiano JJ, Thawy Y, Frame JD. Reconstructive surgery with Integra dermal regeneration template: histologic study, clinical evaluation, and current practice. Plast Reconstr Surg. 2006 Jun;117(7 Suppl):160S-174S. doi: 10.1097/01.prs.0000222609.40461.68. PMID 16799385
- [Background] Wood FM, Giles N, Stevenson A, Rea S, Fear M. Characterisation of the cell suspension harvested from the dermal epidermal junction using a ReCell(R) kit. Burns. 2012 Feb;38(1):44-51. doi: 10.1016/j.burns.2011.03.001. Epub 2011 Nov 12. PMID 22079538
- [Background] Waaijman T, Breetveld M, Ulrich M, Middelkoop E, Scheper RJ, Gibbs S. Use of a collagen-elastin matrix as transport carrier system to transfer proliferating epidermal cells to human dermis in vitro. Cell Transplant. 2010;19(10):1339-48. doi: 10.3727/096368910X507196. Epub 2010 Jun 3. PMID 20525428
- [Background] Wood FM, Stoner ML, Fowler BV, Fear MW. The use of a non-cultured autologous cell suspension and Integra dermal regeneration template to repair full-thickness skin wounds in a porcine model: a one-step process. Burns. 2007 Sep;33(6):693-700. doi: 10.1016/j.burns.2006.10.388. Epub 2007 May 7. PMID 17485177

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ReCell | Control
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Trial closed | 1 | 0

BASELINE CHARACTERISTICS:
Population: did not enroll any additional participants
Groups:
- Total: Total of all reporting groups
Arm/Group | ReCell | Control | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (0) |  | 29 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Event
Description: Number of patients with a treatment-related adverse events requiring surgical intervention prior to Week 12 post-treatment and all serious adverse event (SAE) occurrences throughout the study
Time Frame: Prior to or at 12 weeks
Population: did not enroll any additional participants
Measure: Count of Participants; unit: Participants
Arm/Group | ReCell | Control
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

2. Secondary Outcome: Number of Participants With Confirmed Treatment Area Closure
Description: Complete wound closure is defined as skin wound re-epithelialization at 95% or greater at treated wound site and donor sites confirmed at two consecutive study visits at least 2 weeks apart by direct visualization by a qualified clinician blinded to treatment assignment. The incidence of complete wound closure is hypothesized to be non-inferior for ReCell-treated areas as compared to control areas.
Time Frame: Prior to or at 6 weeks
Population: did not enroll any additional participants
Measure: Count of Participants; unit: Participants
Arm/Group | ReCell | Control
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks and 24 weeks post-operation
Description: Do not differ from clinicaltrials.gov definitions.
Arm/Group | ReCell | Control
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ReCell (N=1) | Control (N=0)
Graft Sloughing (Surgical and medical procedures) | 1 (1) | 0 (0)
Malodorous wound (Surgical and medical procedures) | 1 (1) | 0 (0)
Exudate around graft (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT02469168/Prot_SAP_000.pdf
  • Informed Consent Form (2014-11-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT02469168/ICF_001.pdf